CLINICAL TRIAL: NCT02406118
Title: Phase II Clinical Trial for the Evaluation of the Efficacy of Transanal Total Mesorectal Excision
Brief Title: Phase II Clinical Trial for the Evaluation of the Efficacy of Transanal TME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Dae Kyung Sohn, MD., PHD, Center for Colorectal Cancer, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2015-0033
Record Dates: First submitted 2015-03-25; First posted 2015-04-02 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Rectal Cancer
Keywords: transanal TME quality; CRM
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transanal total mesorectal excision (Experimental): Laparoscopy-assisted transanal total mesorectal excision
  Interventions: Procedure: Transanal total mesorectal excision

INTERVENTIONS:
Procedure: Transanal total mesorectal excision — Subjects will have their rectal cancer removed using a technique combining surgery through the anus and standard laparoscopy. Transanal visualization will be using endoscopy. At the end of the procedure, the rectum will be removed though the anus or ileostomy formation site, the bowel will be re-connected to the anus, and a temporary diverting stoma will be created, which is standard of care following surgery for this type of cancer.
  Other Names: Laparoscopy-assisted transanal TME

SUMMARY:
The purpose of this study is evaluation of the safety and the efficacy of transanal total mesorectal excision.

DETAILED DESCRIPTION:
Subjects will have their rectal cancer removed using a technique combining surgery through the anus and standard laparoscopy. Transanal visualization will be using endoscopy. At the end of the procedure, the rectum will be removed though the anus or ileostomy formation site, the bowel will be re-connected to the anus, and a temporary diverting stoma will be created, which is standard of care following surgery for this type of cancer.

ELIGIBILITY:
Inclusion Criteria:

1. age: 20-80 years
2. biopsy-proven adenocarcinoma of the rectum
3. clinical staging (c or yc): T0-3, N0-2, M0
4. Rectal cancer located 3-12 cm from the anal verge
5. ECOG performance status: 2 or less
6. BMI: less than 30

Exclusion Criteria:

1. Synchronous colon cancer or other malignancy
2. Obstructing rectal cancer
3. Pregnant or breast-feeding
4. Receiving any other study agents
5. Fecal incontinence
6. History of prior colorectal cancer or inflammatory bowel disease
7. Tumor size: more than 7cm in long diameter
8. CRM: mesorectal fascia involvement or less than 1 mm on MRI

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
TME quality & circumferential resection margin (CRM) | the day of trananal TME
  The quality of the mesorectum was determined using pathology reports and scored using three grades:
  * Complete: intact mesorectum with only minor irregularities of a smooth mesorectal surface. No defect is deeper than 5 mm, and there is no coning toward the distal margin of the specimen. There is a smooth circumferential resection margin on slicing.
  * Nearly complete: moderate bulk to the mesorectum, but irregularity of the mesorectal surface. Moderate coning of the specimen is allowed. At no site is the muscularis propria visible, with the exception of the insertion of the levator muscles.
  * Incomplete: little bulk to mesorectum with defects down onto muscularis propria and/or very irregular circumferential resection margin.

SECONDARY OUTCOMES:
30-day postoperative complications | 1 month after surgery
Number of harvested Lymph Nodes | the day of surgery

OTHER OUTCOMES:
2-year local recurrence free survival | 2 years after surgery
5-year overall survival | 5 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dae Kyung Sohn, Principal Investigator — NCC,Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Park SC, Sohn DK, Kim MJ, Chang HJ, Han KS, Hyun JH, Joo J, Oh JH. Phase II Clinical Trial to Evaluate the Efficacy of Transanal Endoscopic Total Mesorectal Excision for Rectal Cancer. Dis Colon Rectum. 2018 May;61(5):554-560. doi: 10.1097/DCR.0000000000001058. PMID 29624549